CLINICAL TRIAL: NCT01250119
Title: Assess the Incidence of Mutations in the Tyrosine Kinase Domain of the Endothelial Growth Factor Receptor in UK Patients With Newly Diagnosed Metastatic or Recurrent Non-small Cell Lung Cancer and to Investigate the Quality of Life of These Patients Undergoing First-line Therapy With Erlotinib.
Brief Title: A Study to Assess the Incidence of EGFR Mutation in Patients With Newly Diagnosed Locally Advanced or Metastatic Non-Small Cell Lung Cancer in the UK, And of Tarceva (Erlotinib) as First-Line Therapy in EGFR Mutation Positive Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25279; 2010-021120-96
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg daily, orally

SUMMARY:
This study will assess the prevalence of epidermal growth factor receptor (EGFR) mutations in newly diagnosed patients with locally advanced or metastatic non-small cell lung cancer (NSCLC). Patients with positive EGFR mutation results will enter an open-label, single arm study to evaluate progression-free survival and quality of life with first-line Tarceva (erlotinib) therapy. Patients will receive Tarceva at a dose of 150 mg orally daily. Anticipated time on study treatment is until progressive disease or unacceptable toxicity occurs. Patients with negative EGFR mutation results will be offered treatment as per the centre's standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Locally advanced or metastatic (stage IIIB/IV) non-small cell lung cancer (NSCLC)
* ECOG performance status 0-3
* Treatment phase: histologically confirmed EGFR exon 19 deletion or exon 21 mutation in the diagnostic phase of the study
* Adequate haematological, liver and renal function
* Female patients must be postmenopausal, surgically sterile, or agree to use a barrier method of contraception
* Male patients must be surgically sterile or agree to use a barrier method of contraception

Exclusion Criteria:

* Previous treatment for NSCLC with chemotherapy or therapy against EGFR, either with antibody or small molecule (tyrosine kinase inhibitor)
* Symptomatic cerebral metastases
* Pregnant or lactating women
* Any other concomitant anti-cancer therapy (until disease progression and discontinuation of Tarceva therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United Kingdom (16):
  - Belfast
  - Bradford
  - Brighton
  - Chelsmford
  - Colchester
  - Dudley
  - Glasgow
  - Grimsby
  - London
  - Newtownards
  - Portadown
  - Rhyl
  - Sutton in Ashfield
  - Truro
  - Westcliffe-on-sea
  - York

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-small-cell Lung Cancer (NSCLC) Group: During the Diagnostic Phase participants newly diagnosed with recurrent or metastatic NSCLC were tested for Epidermal Growth Factor Receptor (EGFR) exon 19 deletions or exon 21 (L858R) mutations.
- Erlotinib 150 Milligrams Per Day (mg/Day): During the Treatment Phase participants found to have a tumour with EGFR exon 19 deletion or exon 21 (L858R) mutations received erlotinib 150 mg/day as a single oral dose until progressive disease (PD), death, unacceptable toxicity or withdrawal of consent.
Period: Diagnostic Phase
Arm/Group | Non-small-cell Lung Cancer (NSCLC) Group | Erlotinib 150 Milligrams Per Day (mg/Day)
Started | 688 | 0
Completed | 575 (Completed refers to participants with both positive and negative EGFR mutation test result.) | 0
Not Completed | 113 | 0
Not completed — Failed to Produce a Test Results | 69 | 0
Not completed — Participants Not Tested | 44 | 0
Period: Treatment Phase
Arm/Group | Non-small-cell Lung Cancer (NSCLC) Group | Erlotinib 150 Milligrams Per Day (mg/Day)
Started | 0 | 41 (Out of 52 participants with positive EGFR mutation test result, only 41 participants were treated.)
Completed | 0 | 0
Not Completed | 0 | 41
Not completed — Progressive Disease | 0 | 32
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Unknown reason | 0 | 4

BASELINE CHARACTERISTICS:
Population: Diagnostic population: All participants newly diagnosed with recurrent or metastatic NSCLC who entered the study and signed the consent form were included in this population.
Groups:
- NSCLC Group: During the Diagnostic Phase participants newly diagnosed with recurrent or metastatic NSCLC were tested for EGFR exon 19 deletions or exon 21 (L858R) mutations.
Arm/Group | NSCLC Group
Number analyzed (Participants) | 688
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299
  Male | 389

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Tested Positive for EGFR Mutations
Description: All participants newly diagnosed with recurrent or metastatic NSCLC were tested for EGFR exon 19 deletion or exon 21 mutations.
Time Frame: 14 days
Population: Diagnostic population; Only participants who were tested for EGFR mutations were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Group
Number analyzed (Participants) | 644
percentage of participants | 8.1

2. Secondary Outcome: Percentage of Participants With a Response by Best Objective Tumor Response
Description: Best objective response was defined as the best response recorded from the start of treatment until disease progression/recurrence. Tumor response was assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1". Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). Partial Response (PR): At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Screening, Day 1 of each 6 week visit starting from Visit 3 until PD, Death, Unacceptable Toxicity or Withdrawal of Consent up to 34 months
Population: Intention-to-treat (ITT) population: All participants in the target population who were eligible for treatment and who actually received one dose of treatment.
Measure: Number; unit: percentage of participants
Groups:
- Erlotinib 150 mg/Day: During the Treatment Phase participants found to have a tumor with EGFR exon 19 deletion or exon 21 (L858R) mutations received erlotinib 150 mg/day as a single oral dose until PD, death, unacceptable toxicity or withdrawal of consent.
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
percentage of participants
  CR | 0.0
  PR | 84.8
  SD | 9.1
  PD | 6.1

3. Primary Outcome: Percentage of Participants With EGFR Mutations by Subgroup
Description: Incidence of EGFR mutations were summarized with respect to different subgroups as follows: (1) equals (=) Histopathology, (2) = Stage of disease, (3) = Age at consent, (4) = Gender, (5) = Race, (6) = Smoking history.
Time Frame: 14 Days
Population: Only participants with a valid EGFR mutations test result were included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- EGFR Positive: All participants who tested positive for EGFR mutations were included in this group.
- EGFR Negative: All participants who tested negative for EGFR mutations were included in this group.
Arm/Group | EGFR Positive | EGFR Negative
Number analyzed (Participants) | 52 | 523
percentage of participants
  (1) Squamous cell carcinoma | 0.0 | 22.6
  (1) Adenocarcinoma | 100.0 | 67.3
  (1) Bronchoalveolar carcinoma | 0 | 1.7
  (1) Large cell carcinoma | 0 | 0.6
  (1) Other | 0 | 7.8
  (2) Unresectable Stage IIIB | 1.9 | 11.9
  (2) Stage IIIB with malignant effusions | 1.9 | 3.4
  (2) Stage IV | 96.2 | 84.7
  (3) Less than 70 years | 73.1 | 55.6
  (3) Greater than 70 years | 26.9 | 44.4
  (4) Male | 23.1 | 60.8
  (4) Female | 76.9 | 39.2
  (5) Asian | 13.5 | 2.9
  (5) Black | 9.6 | 3.3
  (5) Caucasian | 75.0 | 93.5
  (5) Other | 1.9 | 0.4
  (6) Never smoked | 44.2 | 7.8
  (6) Previous smoker | 44.2 | 60.6
  (6) Current smoker | 7.7 | 31.0
  (6) Missing | 3.8 | 0.6
Statistical Analysis 1: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0000, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for histopathology; Univariate analysis
Statistical Analysis 2: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.1038, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for histopathology; Multivariate analysis (6 main effects only)
Statistical Analysis 3: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0588, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for stage of disease; Univariate analysis
Statistical Analysis 4: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.4802, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for stage of disease; Multivariate analysis (6 main effects only)
Statistical Analysis 5: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0147, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for age at consent; Multivariate analysis (6 main effects only)
Statistical Analysis 6: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.1181, Wald Test; [statistical method as in outcome 3, analysis 5]
Statistical Analysis 7: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0000, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for gender; Univariate analysis
Statistical Analysis 8: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0006, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for gender; Multivariate analysis (6 main effects only)
Statistical Analysis 9: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0004, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for race; Univariate analysis
Statistical Analysis 10: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.3371, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for race; Multivariate analysis (6 main effects only)
Statistical Analysis 11: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0000, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for smoking history; Univariate analysis
Statistical Analysis 12: Comparison: EGFR Positive vs EGFR Negative; Test type: Superiority or Other; p = 0.0001, Wald Test; Test for difference in incidence of EGFR mutations for each subgroup controlled for smoking history; Multivariate analysis (6 main effects only)

4. Secondary Outcome: Probability of Being Alive and Free of Progression by Timepoint
Description: Progression Free Survival (PFS) was defined as the interval (number of days) from the trial treatment start date to the earlier of the date of the first tumor response assessment of PD or the date of death by any cause. Participants who experienced neither of these events or who were lost to followup at the time of the analysis were censored at date of last contact. PFS was summarized according to the Kaplan-Meier method.
Time Frame: Months 0, 3, 6, 9, 12, 15, and 18
Population: ITT population
Measure: Number (95% Confidence Interval); unit: probability of being alive
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
probability of being alive
  0 Months | 1.00 [1.00 to 1.00]
  3 Months | 0.97 [0.81 to 1.00]
  6 Months | 0.94 [0.78 to 0.98]
  9 Months | 0.73 [0.54 to 0.85]
  12 Months | 0.54 [0.36 to 0.69]
  15 Months | 0.37 [0.21 to 0.54]
  18 Months | 0.22 [0.09 to 0.39]

5. Secondary Outcome: Survival Time in Months
Description: Duration of time in months from Screening until Death due to any cause.
Time Frame: Baseline, Day 1 of each 6-week visit starting from Visit 3 until PD, Death, Unacceptable toxicity or Withdrawal of consent up to 34 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
months | 12.57 [10.10 to 16.53]

6. Secondary Outcome: Quality of Life Assessment Using EuroQol(EQ) 5D Visual Analog Score (VAS) Instrument
Description: The EQ-5D contains a descriptive system that measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The EQ-5D also contains a visual analog scale (EQ-VAS), which records the respondent's self-rated health status on a vertical graduated visual analog scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). A negative change indicates improvement.
Time Frame: Screening, Baseline and Final or Withdrawal Visit up to 34 months
Population: ITT population; number (n) = number of participants analyzed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 40
mm
  Screening (n=40) | 62.6 (23.5)
  Baseline (n=20) | 65.4 (19.9)
  Final visit/Withdrawal (n=20) | 63.0 (22.4)
  Change from Baseline Final visit(n=20) | -0.4 (22.0)

7. Secondary Outcome: Percentage of Participants With Problems With Mobility as Assessed Using the EQ-5D
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The participants were required to rate their mobility as the following categories: Category 1. I have no problems in walking about; Category 2. I have some problems in walking about; Category 3. I am confined to bed.
Time Frame: Baseline (Visit 1), Days 10 to 14 (Visit 2), Day 1 of every 6 weeks until PD, Death, Unacceptable toxicity or Withdrawal of consent up to 34 months
Population: ITT population; n = number of participants analyzed at for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
percentage of participants
  Screening Category 1 (n=41) | 43.9
  Screening Category 2 (n=41) | 56.1
  Screening Category 3 (n=41) | 0.0
  Visit 01 Category 1 (n=20) | 45.0
  Visit 01 Category 2 (n=20) | 55.0
  Visit 01 Category 3 (n=20) | 0.0
  Visit 02 Category 1 (n=33) | 45.5
  Visit 02 Category 2 (n=33) | 54.5
  Visit 02 Category 3 (n=33) | 0.0
  Visit 03 Category 1 (n=30) | 56.7
  Visit 03 Category 2 (n=30) | 43.3
  Visit 03 Category 3 (n=30) | 0.0
  Visit 04 Category 1 (n=29) | 51.7
  Visit 04 Category 2 (n=29) | 48.3
  Visit 04 Category 3 (n=29) | 0.0
  Visit 05 Category 1 (n=33) | 54.5
  Visit 05 Category 2 (n=33) | 45.5
  Visit 05 Category 3 (n=33) | 0.0
  Visit 06 Category 1 (n=31) | 54.8
  Visit 06 Category 2 (n=31) | 45.2
  Visit 06 Category 3 (n=31) | 0.0
  Visit 07 Category 1 (n=29) | 58.6
  Visit 07 Category 2 (n=29) | 41.4
  Visit 07 Category 3 (n=29) | 0.0
  Visit 08 Category 1 (n=27) | 55.6
  Visit 08 Category 2 (n=27) | 44.4
  Visit 08 Category 3 (n=27) | 0.0
  Visit 09 Category 1 (n=24) | 62.5
  Visit 09 Category 2 (n=24) | 37.5
  Visit 09 Category 3 (n=24) | 0.0
  Visit 10 Category 1 (n=21) | 42.9
  Visit 10 Category 2 (n=21) | 57.1
  Visit 10 Category 3 (n=21) | 0.0
  Visit 11 Category 1 (n=13) | 46.2
  Visit 11 Category 2 (n=13) | 53.8
  Visit 11 Category 3 (n=13) | 0.0
  Visit 12 Category 1 (n=11) | 45.5
  Visit 12 Category 2 (n=11) | 54.5
  Visit 12 Category 3 (n=11) | 0.0
  Visit 13 Category 1 (n=9) | 55.6
  Visit 13 Category 2 (n=9) | 44.4
  Visit 13 Category 3 (n=9) | 0.0
  Visit 14 Category 1 (n=8) | 50.0
  Visit 14 Category 2 (n=8) | 50.0
  Visit 14 Category 3 (n=8) | 0.0
  Visit 15 Category 1 (n=5) | 40.0
  Visit 15 Category 2 (n=5) | 60.0
  Visit 15 Category 3 (n=5) | 0.0
  Visit 16 Category 1 (n=4) | 25.0
  Visit 16 Category 2 (n=4) | 75.0
  Visit 16 Category 3 (n=4) | 0.0
  Visit 17 Category 1 (n=4) | 25.0
  Visit 17 Category 2 (n=4) | 75.0
  Visit 17 Category 3 (n=4) | 0.0
  Visit 18 Category 1 (n=3) | 33.3
  Visit 18 Category 2 (n=3) | 66.7
  Visit 18 Category 3 (n=3) | 0.0
  Visit 19 Category 1 (n=2) | 50.0
  Visit 19 Category 2 (n=2) | 50.0
  Visit 19 Category 3 (n=2) | 0.0
  Visit 20 Category 1 (n=2) | 50.0
  Visit 20 Category 2 (n=2) | 50.0
  Visit 20 Category 3 (n=2) | 0.0
  Visit 21 Category 1 (n=2) | 50.0
  Visit 21 Category 2 (n=2) | 50.0
  Visit 21 Category 3 (n=2) | 0.0
  Visit 22 Category 1 (n=1) | 0.0
  Visit 22 Category 2 (n=1) | 100.0
  Visit 22 Category 3 (n=1) | 0.0
  Visit 23 Category 1 (n=1) | 0.0
  Visit 23 Category 2 (n=1) | 100.0
  Visit 23 Category 3 (n=1) | 0.0
  Visit 24 Category 1 (n=1) | 0.0
  Visit 24 Category 2 (n=1) | 100.0
  Visit 24 Category 3 (n=1) | 0.0
  Visit 25 Category 1 (n=1) | 0.0
  Visit 25 Category 2 (n=1) | 100.0
  Visit 25 Category 3 (n=1) | 0.0
  Final visit/Withdraw Category 1 (n=21) | 33.3
  Final visit/Withdraw Category 2 (n=21) | 66.7
  Final visit/Withdraw Category 3 (n=21) | 0.0

8. Secondary Outcome: Percentage of Participants With Problems With Self-Care as Assessed Using the EQ-5D
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The participants were required to rate their self-care as the following categories: Category 1. I have no problems with self-care; Category 2. I have some problems washing or dressing myself; Category 3. I am unable to wash or dress myself.
Time Frame: as for outcome 7
Population: ITT population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
percentage of participants
  Screening Category 1 (n=41) | 78.0
  Screening Category 2 (n=41) | 17.1
  Screening Category 3 (n=41) | 4.9
  Visit 01 Category 1 (n=20) | 80.0
  Visit 01 Category 2 (n=20) | 20.0
  Visit 01 Category 3 (n=20) | 0.0
  Visit 02 Category 1 (n=33) | 81.8
  Visit 02 Category 2 (n=33) | 18.2
  Visit 02 Category 3 (n=33) | 0.0
  Visit 03 Category 1 (n=29) | 86.2
  Visit 03 Category 2 (n=29) | 13.8
  Visit 03 Category 3 (n=29) | 0.0
  Visit 04 Category 1 (n=28) | 82.1
  Visit 04 Category 2 (n=28) | 17.9
  Visit 04 Category 3 (n=28) | 0.0
  Visit 05 Category 1 (n=33) | 78.8
  Visit 05 Category 2 (n=33) | 21.2
  Visit 05 Category 3 (n=33) | 0.0
  Visit 06 Category 1 (n=31) | 83.9
  Visit 06 Category 2 (n=31) | 16.1
  Visit 06 Category 3 (n=31) | 0.0
  Visit 07 Category 1 (n=29) | 79.3
  Visit 07 Category 2 (n=29) | 20.7
  Visit 07 Category 3 (n=29) | 0.0
  Visit 08 Category 1 Visit 08 Category 1 (n=27) | 85.2
  Visit 08 Category 2 (n=27) | 14.8
  Visit 08 - Category 3 (n=27) | 0.0
  Visit 09 Category 1 (n=24) | 75.0
  Visit 09 Category 2 (n=24) | 25.0
  Visit 09 Category 3 (n=24) | 0.0
  Visit 10 Category 1 (n=21) | 71.4
  Visit 10 Category 2 (n=21) | 28.6
  Visit 10 Category 3 (n=21) | 0.0
  Visit 11 Category 1 (n=13) | 61.5
  Visit 11 Category 2 (n=13) | 38.5
  Visit 11 Category 3 (n=13) | 0.0
  Visit 12 Category 1 (n=11) | 54.5
  Visit 12 Category 2 (n=11) | 45.5
  Visit 12 Category 3 (n=11) | 0.0
  Visit 13 Category 1 (n=9) | 55.6
  Visit 13 Category 2 (n=9) | 44.4
  Visit 13 Category 3 (n=9) | 0.0
  Visit 14 Category 1 (n=8) | 62.5
  Visit 14 Category 2 (n=8) | 37.5
  Visit 14 Category 3 (n=8) | 0.0
  Visit 15 Category 1 (n=5) | 40.0
  Visit 15 Category 2 (n=5) | 60.0
  Visit 15 Category 3 (n=5) | 0.0
  Visit 16 Category 1 (n=4) | 50.0
  Visit 16 Category 2 ((n=4)) | 50.0
  Visit 16 Category 3 (n=4) | 0.0
  Visit 17 Category 1 (n=4) | 50.0
  Visit 17 Category 2 (n=4) | 50.0
  Visit 17 Category 3 (n=4) | 0.0
  Visit 18 Category 1 (n=3) | 33.3
  Visit 18 Category 2 (n=3) | 66.7
  Visit 18 Category 3 (n=3) | 0.0
  Visit 19 Category 1 (n=2) | 50.0
  Visit 19 Category 2 (n=2) | 50.0
  Visit 19 Category 3 (n=2) | 0.0
  Visit 20 Category 1 (n=2) | 50.0
  Visit 20 Category 2 (n=2) | 50.0
  Visit 20 Category 3 (n=2) | 0.0
  Visit 21 Category 1 (n=2) | 50.0
  Visit 21 Category 2 (n=2) | 50.0
  Visit 21 Category 3 (n=2) | 0.0
  Visit 22 Category 1 (n=1) | 100.0
  Visit 22 Category 2 (n=1) | 0.0
  Visit 22 Category 3 (n=1) | 0.0
  Visit 23 Category 1 (n=1) | 0.0
  Visit 23 Category 2 (n=1) | 100.0
  Visit 23 Category 3 (n=1) | 0.0
  Visit 24 Category 1 (n=1) | 0.0
  Visit 24 Category 2 (n=1) | 100.0
  Visit 24 Category 3 (n=1) | 0.0
  Visit 25 Category 1 (n=1) | 0.0
  Visit 25 Category 2 (n=1) | 100.0
  Visit 25 Category 3 (n=1) | 0.0
  Final visit/Withdraw Category 1 (n=21) | 66.7
  Final visit/Withdraw Category 2 (n=21) | 33.3
  Final visit/Withdraw Category 3 (n=21) | 0.0

9. Secondary Outcome: Percentage of Participants With Problems With Usual Activities as Assessed Using the EQ-5D
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The participants were required to rate their ability to perform usual activities as the following categories: Category 1. I have no problems with performing my usual activities; Category 2. I have some problems with performing my usual activities; Category 3. I am unable to perform my usual activities.
Time Frame: as for outcome 7
Population: ITT population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
percentage of participants
  Screening Category 1 (n=41) | 39.0
  Screening Category 2 (n=41) | 46.3
  Screening Category 3 (n=41) | 14.6
  Visit 01 Category 1 (n=20) | 40.0
  Visit 01 Category 2 (n=20) | 50.0
  Visit 01 Category 3 (n=20) | 10.0
  Visit 02 Category 1 (n=33) | 36.4
  Visit 02 Category 2 (n=33) | 60.6
  Visit 02 Category 3 (n=33) | 3.0
  Visit 03 Category 1 (n=30) | 40.0
  Visit 03 Category 2 (n=30) | 53.3
  Visit 03 Category 3 (n=30) | 6.7
  Visit 04 Category 1 (n=29) | 51.7
  Visit 04 Category 2 (n=29) | 44.8
  Visit 04 Category 3 (n=29) | 3.4
  Visit 05 Category 1 (n=33) | 51.5
  Visit 05 Category 2 (n=33) | 48.5
  Visit 05 Category 3 (n=33) | 0.0
  Visit 06 Category 1 (n=31) | 45.2
  Visit 06 Category 2 (n=31) | 54.8
  Visit 06 Category 3 (n=31) | 0.0
  Visit 07 Category 1 (n=29) | 48.3
  Visit 07 Category 2 (n=29) | 51.7
  Visit 07 Category 3 (n=29) | 0.0
  Visit 08 Category 1 (n=27) | 40.7
  Visit 08 Category 2 (n=27) | 59.3
  Visit 08 Category 3 (n=27) | 0.0
  Visit 09 Category 1 (n=24) | 33.3
  Visit 09 Category 2 (n=24) | 66.7
  Visit 09 Category 3 (n=24) | 0.0
  Visit 10 Category 1 (n=21) | 38.1
  Visit 10 Category 2 (n=21) | 61.9
  Visit 10 Category 3 (n=21) | 0.0
  Visit 11 Category 1 (n=13) | 30.8
  Visit 11 Category 2 (n=13) | 69.2
  Visit 11 Category 3 (n=13) | 0.0
  Visit 12 Category 1 (n=11) | 27.3
  Visit 12 Category 2 (n=11) | 72.7
  Visit 12 Category 3 (n=11) | 0.0
  Visit 13 Category 1 (n=9) | 22.2
  Visit 13 Category 2 (n=9) | 77.8
  Visit 13 Category 3 (n=9) | 0.0
  Visit 14 Category 1 (n=8) | 37.5
  Visit 14 Category 2 (n=8) | 62.5
  Visit 14 Category 3 (n=8) | 0.0
  Visit 15 Category 1 (n=5) | 20.0
  Visit 15 Category 2 (n=5) | 80.0
  Visit 15 Category 3 (n=5) | 0.0
  Visit 16 Category 1 (n=4) | 25.0
  Visit 16 Category 2 (n=4) | 75.0
  Visit 16 Category 3 (n=4) | 0.0
  Visit 17 Category 1 (n=4) | 25.0
  Visit 17 Category 2 (n=4) | 75.0
  Visit 17 Category 3 (n=4) | 0.0
  Visit 18 Category 1 (n=3) | 33.3
  Visit 18 Category 2 (n=3) | 66.7
  Visit 18 Category 3 (n=3) | 0.0
  Visit 19 Category 1 (n=2) | 50.0
  Visit 19 Category 2 (n=2) | 50.0
  Visit 19 Category 3 (n=2) | 0.0
  Visit 20 Category 1 (n=2) | 50.0
  Visit 20 Category 2 (n=2) | 50.0
  Visit 20 Category 3 (n=2) | 0.0
  Visit 21 Category 1 (n=2) | 50.0
  Visit 21 Category 2 (n=2) | 50.0
  Visit 21 Category 3 (n=2) | 0.0
  Visit 22 Category 1 (n=1) | 0.0
  Visit 22 Category 2 (n=1) | 100.0
  Visit 22 Category 3 (n=1) | 0.0
  Visit 23 Category 1 (n=1) | 0.0
  Visit 23 Category 2 (n=1) | 100.0
  Visit 23 Category 3 (n=1) | 0.0
  Visit 24 Category 1 (n=1) | 0.0
  Visit 24 Category 2 (n=1) | 100.0
  Visit 24 Category 3 (n=1) | 0.0
  Visit 25 Category 1 (n=1) | 0.0
  Visit 25 Category 2 (n=1) | 100.0
  Visit 25 Category 3 (n=1) | 0.0
  Final visit/Withdrawal Category 1 (n=21) | 33.3
  Final visit/Withdrawal Category 2 (n=21) | 61.9
  Final visit/Withdrawal Category 3 (n=21) | 4.8

10. Secondary Outcome: Percentage of Participants With Pain/Discomfort as Assessed Using the EQ-5D
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The participants were required to rate their pain as the following categories: Category 1. I have no pain or discomfort; Category 2. I have moderate pain or discomfort; Category 3. I have extreme pain or discomfort.
Time Frame: as for outcome 7
Population: ITT population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
percentage of participants
  Screening Category 1 (n=41) | 29.3
  Screening Category 2 (n=41) | 63.4
  Screening Category 3 (n=41) | 7.3
  Visit 01 Category 1 (n=20) | 10.0
  Visit 01 Category 2 (n=20) | 85.0
  Visit 01 Category 3 (n=20) | 5.0
  Visit 02 Category 1 (n=32) | 43.8
  Visit 02 Category 2 (n=32) | 56.3
  Visit 02 Category 3 (n=32) | 0.0
  Visit 03 Category 1 (n=30) | 40.0
  Visit 03 Category 2 (n=30) | 60.0
  Visit 03 Category 3 (n=30) | 0.0
  Visit 04 Category 1 (n=29) | 55.2
  Visit 04 Category 2 (n=29) | 37.9
  Visit 04 Category 3 (n=29) | 6.9
  Visit 05 Category 1 (n=33) | 45.5
  Visit 05 Category 2 (n=33) | 51.5
  Visit 05 Category 3 (n=33) | 3.0
  Visit 06 Category 1 (n=31) | 48.4
  Visit 06 Category 2 (n=31) | 51.6
  Visit 06 Category 3 (n=31) | 0.0
  Visit 07 Category 1 (n=29) | 48.3
  Visit 07 Category 2 (n=29) | 51.7
  Visit 07 Category 3 (n=29) | 0.0
  Visit 08 Category 1 (n=27) | 37.0
  Visit 08 Category 2 (n=27) | 59.3
  Visit 08 Category 3 (n=27) | 3.7
  Visit 09 Category 1 (n=24) | 50.0
  Visit 09 Category 2 (n=24) | 37.5
  Visit 09 Category 3 (n=24) | 12.5
  Visit 10 Category 1 (n=21) | 42.9
  Visit 10 Category 2 (n=21) | 47.6
  Visit 10 Category 3 (n=21) | 9.5
  Visit 11 Category 1 (n=13) | 46.2
  Visit 11 Category 2 (n=13) | 53.8
  Visit 11 Category 3 (n=13) | 0.0
  Visit 12 Category 1 (n=11) | 45.5
  Visit 12 Category 2 (n=11) | 36.4
  Visit 12 Category 3 (n=11) | 18.2
  Visit 13 Category 1 (n=9) | 44.4
  Visit 13 Category 2 (n=9) | 55.6
  Visit 13 Category 3 (n=9) | 0.0
  Visit 14 Category 1 (n=8) | 62.5
  Visit 14 Category 2 (n=8) | 37.5
  Visit 14 Category 3 (n=8) | 0.0
  Visit 15 Category 1 (n=5) | 60.0
  Visit 15 Category 2 (n=5) | 40.0
  Visit 15 Category 3 (n=5) | 0.0
  Visit 16 Category 1 (n=4) | 25.0
  Visit 16 Category 2 (n=4) | 75.0
  Visit 16 Category 3 (n=4) | 0.0
  Visit 17 Category 1 (n=4) | 25.0
  Visit 17 Category 2 (n=4) | 75.0
  Visit 17 Category 3 (n=4) | 0.0
  Visit 18 Category 1 (n=3) | 0.0
  Visit 18 Category 2 (n=3) | 100.0
  Visit 18 Category 3 (n=3) | 0.0
  Visit 19 Category 1 (n=2) | 0.0
  Visit 19 Category 2 (n=2) | 100.0
  Visit 19 Category 3 (n=2) | 0.0
  Visit 20 Category 1 (n=2) | 0.0
  Visit 20 Category 2 (n=2) | 100.0
  Visit 20 Category 3 (n=2) | 0.0
  Visit 21 Category 1 (n=2) | 0.0
  Visit 21 Category 2 (n=2) | 100.0
  Visit 21 Category 3 (n=2) | 0.0
  Visit 22 Category 1 (n=1) | 100.0
  Visit 22 Category 2 (n=1) | 0.0
  Visit 22 Category 3 (n=1) | 0.0
  Visit 23 Category 1 (n=1) | 0.0
  Visit 23 Category 2 (n=1) | 100.0
  Visit 23 Category 3 (n=1) | 0.0
  Visit 24 Category 1 (n=1) | 0.0
  Visit 24 Category 2 (n=1) | 100.0
  Visit 24 Category 3 (n=1) | 0.0
  Visit 25 Category 1 (n=1) | 0.0
  Visit 25 Category 2 (n=1) | 100.0
  Visit 25 Category 3 (n=1) | 0.0
  Final visit/Withdrawal Category 1 (n=21) | 38.1
  Final visit/Withdrawal Category 2 (n=21) | 57.1
  Final visit/Withdrawal Category 3 (n=21) | 4.8

11. Secondary Outcome: Percentage of Participants With Anxiety/Depression as Assessed Using the EQ-5D
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The participants were required to rate their pain as the following categories: Category 1. I am not anxious or depressed; Category 2. I am moderately anxious or depressed; Category 3.I am extremely anxious or depressed.
Time Frame: as for outcome 7
Population: ITT population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 41
percentage of participants
  Screening Category 1 (n=40) | 52.5
  Screening Category 2 (n=40) | 37.5
  Screening Category 3 (n=40) | 10.0
  Visit 01 Category 1 (n=19) | 57.9
  Visit 01 Category 2 (n=19) | 42.1
  Visit 01 Category 3 (n=19) | 0.0
  Visit 02 Category 1 (n=33) | 57.6
  Visit 02 Category 2 (n=33) | 42.4
  Visit 02 Category 3 (n=33) | 0.0
  Visit 03 Category 1 (n=30) | 43.3
  Visit 03 Category 2 (n=30) | 56.7
  Visit 03 Category 3 (n=30) | 0.0
  Visit 04 Category 1 (n=29) | 58.6
  Visit 04 Category 2 (n=29) | 41.4
  Visit 04 Category 3 (n=29) | 0.0
  Visit 05 Category 1 (n=33) | 60.6
  Visit 05 Category 2 (n=33) | 36.4
  Visit 05 Category 3 (n=33) | 3.0
  Visit 06 Category 1 (n=31) | 48.4
  Visit 06 Category 2 (n=31) | 51.6
  Visit 06 Category 3 (n=31) | 0.0
  Visit 07 Category 1 (n=29) | 62.1
  Visit 07 Category 2 (n=29) | 37.9
  Visit 07 Category 3 (n=29) | 0.0
  Visit 08 Category 1 (n=27) | 55.6
  Visit 08 Category 2 (n=27) | 44.4
  Visit 08 Category 3 (n=27) | 0.0
  Visit 09 Category 1 (n=24) | 62.5
  Visit 09 Category 2 (n=24) | 25.0
  Visit 09 Category 3 (n=24) | 12.5
  Visit 10 Category 1 (n=21) | 61.9
  Visit 10 Category 2 (n=21) | 28.6
  Visit 10 Category 3 (n=21) | 9.5
  Visit 11 Category 1 (n=13) | 61.5
  Visit 11 Category 2 (n=13) | 30.8
  Visit 11 Category 3 (n=13) | 7.7
  Visit 12 Category 1 (n=11) | 45.5
  Visit 12 Category 2 (n=11) | 45.5
  Visit 12 Category 3 (n=11) | 9.1
  Visit 13 Category 1 (n=9) | 77.8
  Visit 13 Category 2 (n=9) | 22.2
  Visit 13 Category 3 (n=9) | 0.0
  Visit 14 Category 1 (n=8) | 75.0
  Visit 14 Category 2 (n=8) | 25.0
  Visit 14 Category 3 (n=8) | 0.0
  Visit 15 Category 1 (n=5) | 60.0
  Visit 15 Category 2 (n=5) | 40.0
  Visit 15 Category 3 (n=5) | 0.0
  Visit 16 Category 1 (n=4) | 75.0
  Visit 16 Category 2 (n=4) | 25.0
  Visit 16 Category 3 (n=4) | 0.0
  Visit 17 Category 1 (n=4) | 75.0
  Visit 17 Category 2 (n=4) | 25.0
  Visit 17 Category 3 (n=4) | 0.0
  Visit 18 Category 1 (n=3) | 66.7
  Visit 18 Category 2 (n=3) | 33.3
  Visit 18 Category 3 (n=3) | 0.0
  Visit 19 Category 1 (n=2) | 50.0
  Visit 19 Category 2 (n=2) | 50.0
  Visit 19 Category 3 (n=2) | 0.0
  Visit 20 Category 1 (n=2) | 50.0
  Visit 20 Category 2 (n=2) | 50.0
  Visit 20 Category 3 (n=2) | 0.0
  Visit 21 Category 1 (n=2) | 50.0
  Visit 21 Category 2 (n=2) | 50.0
  Visit 21 Category 3 (n=2) | 0.0
  Visit 22 Category 1 (n=1) | 100.0
  Visit 22 Category 2 (n=1) | 0.0
  Visit 22 Category 3 (n=1) | 0.0
  Visit 23 Category 1 (n=1) | 0.0
  Visit 23 Category 2 (n=1) | 100.0
  Visit 23 Category 3 (n=1) | 0.0
  Visit 24 Category 1 (n=1) | 0.0
  Visit 24 Category 2 (n=1) | 100.0
  Visit 24 Category 3 (n=1) | 0.0
  Visit 25 Category 1 (n=1) | 0.0
  Visit 25 Category 2 (n=1) | 100.0
  Visit 25 Category 3 (n=1) | 0.0
  Final visit/Withdrawal Category 1 (n=21) | 57.1
  Final visit/Withdrawal Category 2 (n=21) | 38.1
  Final visit/Withdrawal Category 3 (n=21) | 4.8

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from Visit 1 (Baseline) until 30 days after the Final/Withdrawal Visit.
Arm/Group | Erlotinib 150 mg/Day
Serious Adverse Events (participants affected / at risk) | 16/41
Other Adverse Events (participants affected / at risk) | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg/Day (N=41)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg/Day (N=41)
Anaemia (Blood and lymphatic system disorders) | 7
Conjunctivitis (Eye disorders) | 3
Dry eye (Eye disorders) | 3
Vision blurred (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 26
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Oral pain (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 4
Chest pain (General disorders) | 3
Fatigue (General disorders) | 14
Mucosal inflammation (General disorders) | 6
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 3
Cellulitis (Infections and infestations) | 3
Lower respiratory tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 4
Paronychia (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 3
Pulmonary function test decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 26
Skin ulcer (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.